CLINICAL TRIAL: NCT06794996
Title: A Phase 2b, Open-label Study to Evaluate the Efficacy and Safety of Inaxaplin in Subjects With Proteinuric APOL1-mediated Kidney Disease With or Without Comorbidities That May Independently Contribute to Chronic Kidney Disease
Brief Title: Inaxaplin in Participants With Proteinuric APOL1 Mediated Kidney Disease With or Without Comorbidities
Acronym: AMPLIFIED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-147-202
Record Dates: First submitted 2025-01-23; First posted 2025-01-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Proteinuric Kidney Disease
Keywords: APOL1-mediated kidney disease (AMKD)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IXP (Inaxaplin) (Experimental): Participants with proteinuric APOL1-mediated kidney disease (AMKD) with or without the comorbidity of Type 2 diabetes mellitus (T2DM) will receive a single dose of IXP once daily, for 13 weeks.
  Interventions: Drug: Inaxaplin

INTERVENTIONS:
Drug: Inaxaplin — Tablets for Oral Administration.
  Other Names: IXP; VX-147

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, and tolerability of Inaxaplin (IXP) in participants with proteinuric APOL1- mediated kidney disease (AMKD).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has an APOL1 genotype of G1/G1, G2/G2, or G1/G2 obtained with a Vertex designated investigational clinical study assay
* Estimated Glomerular Filtration Rate (eGFR) of greater than or equal to (≥) 25 milliliter per minute (mL/min)/1.73m^2 at screening

Key Exclusion Criteria:

* Evidence of Focal Segmental Glomerulosclerosis (FSGS) with a known cause other than due to APOL1 risk variants
* Uncontrolled hypertension

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Urine Albumin-Creatinine Ratio (UACR) | Baseline and At Week 13

SECONDARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline Up To Week 17

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Foundation for Sickle Cell Disease Research, LLC, Hollywood, Florida
  - South Florida Research Institute, Lauderdale Lakes, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Renal Associates, LLC, Columbus, Georgia
  - Georgia Nephrology - Decatur, Decatur, Georgia
  - Javara Inc./Privia Medical Group Georgia, LLC - Fayetteville, Fayetteville, Georgia
  - Georgia Nephrology, Lawrenceville, Georgia
  - Javara Inc. /Privia Medical Group Georgia, LLC - Savannah, Savannah, Georgia
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - LCMC Health, Metairie, Louisiana
  - Ochsner Medical Center - New Orleans - Nephrology, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, LLC - Shreveport, Shreveport, Louisiana
  - Javara Inc./Privia Medical Group, LLC MidAtlantic-Silver Spring, MD, Silver Spring, Maryland
  - Nephrology Associates, P.C., Columbus, Mississippi
  - Nephrology and Hypertension Associates, LTD, Tupelo, Mississippi
  - DaVita Clinical Research, Las Vegas, Nevada
  - Saint Michael's Medical Center - Peter Ho Memorial Clinic, Newark, New Jersey
  - Rutgers Doctors Office Center, Newark, New Jersey
  - Scott Research, Inc., Laurelton, New York
  - NYC Health + Hospital/Harlem, New York, New York
  - North Carolina Nephrology P.A. - Cary Office, Cary, North Carolina
  - UNC Clinical and Translational Research Center, Chapel Hill, North Carolina
  - Duke University Hospital - Children's Health Center, Durham, North Carolina
  - Eastern Nephrology Associates - New Bern Office, New Bern, North Carolina
  - Lewis Katz School of Medicine at Temple University - Section of Nephrology, Philadelphia, Pennsylvania
  - Columbia Nephrology Associates, PA, Columbia, South Carolina
  - Carolina Nephrology, PA, Spartanburg, South Carolina
  - Dallas Renal Group - 2, Dallas, Texas
  - Dallas Renal Group - 1, Dallas, Texas
  - Dallas Nephrology Associates - Dallas Landry Office, Dallas, Texas
  - UTSW Medical Center - Nephrology, Dallas, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - Tks Research, P.L.L.C., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/